CLINICAL TRIAL: NCT02025829
Title: The Role of IL-17 Neutrophils in CF Lung Inflammation
Brief Title: IL-17 Neutrophils in CF Lung Inflammation
Status: Completed | Type: Observational
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: Case Western Reserve University (Other)
Responsible Party: Principal Investigator, James F. Chmiel, Associate Professor of Pediatrics, University Hospitals Cleveland Medical Center
Other Study IDs: 01CH2013
Record Dates: First submitted 2013-12-18; First posted 2014-01-01 (Estimated); Results first posted 2017-03-24 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-01

CONDITIONS: Cystic Fibrosis
Keywords: cystic fibrosis; IL-17 neutrophils
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — peripheral white cells, serum, sputum white cells, sputum supernatants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Clinically Stable: Patients with cystic fibrosis and are clinically stable, 10 subjects with one copy of F508del and 4 subjects with at least one copy of G551D
- Exacerbation: Patients with cystic fibrosis admitted for treatment of a pulmonary exacerbation with IV antibiotics, 10 subjects with one copy of F508del

SUMMARY:
The purpose of this study is to determine whether IL-17 polymorphonuclear leukocytes (PMNs) are central to the disease pathology in CF. This will be determined by demonstrating that IL-17 PMNs are present in the CF airway, correlate with lung function measures, and decrease in patients being treated with IV antibiotics for a pulmonary exacerbation.

DETAILED DESCRIPTION:
This study consists of two parts which will be conducted in parallel. In the first part of the study, 14 subjects will be recruited for the Clinically Stable Cohort. Subjects will be asked to provide 1 gm of expectorated sputum and 40-ml of blood. A cell count and differential will be performed on the sputum followed by analysis for IL-17 PMNs by fluorescence-activated cell sorter (FACS). IL-17 PMNs also will be isolated by running the remainder of the cell pellet through a column of magnetic beads designed for this purpose. These neutrophils will be lysed and intracellular cytokines determined. Sputum supernatants will be stored frozen until analyzed for the presence of IL-1β, IL-6, IL-8, IL-17A, TGF-β, TNF-α, and neutrophil elastase. Clinical data will be captured from the subject's clinical outpatient visit including lung function measures and clinical culture results. IL-17 PMNs will be correlated with lung function measures and inflammatory mediators at baseline.

In the second part of this study, 10 subjects will be recruited for the Exacerbation Cohort. Subjects will provide at least 1 gram of expectorated sputum and 40-ml of blood within 72 hours of hospital admission. Sputum and blood will be processed and analyzed as described above. Sputum and blood also will be obtained at the end of treatment (within 72 hours of completion of IV antibiotics) when the subject is at his or her baseline as determined by the managing physician. Clinical data will be captured from the subject's hospitalization records including lung function measures and clinical culture results.

ELIGIBILITY:
Inclusion Criteria:

* For Both Cohorts: ≥ 18 < 50 years of age
* For Both Cohorts: Must have a documented diagnosis of CF (positive sweat chloride ≥60 milliequivalents (mEq)/liter, by pilocarpine iontophoresis) and/or a genotype with two identifiable mutations consistent with CF accompanied by one or more clinical features with the CF) phenotype
* For Both Cohorts: Chronically infected with P. aeruginosa defined by 2 positive cultures in the past year or 3 in the last two years
* For Both Cohorts: Ability to expectorate mucus
* For Both Cohorts: Ability to provide written informed consent
* For Clinically Stable Cohort: 4 subjects with one copy of G551D
* For Clinically Stable Cohort: 10 subjects who do not have G551D, they must have one copy of F508del
* For Clinically Stable Cohort: CF subjects must have a baseline FEV1 percent predicted > 50% (in the last year, obtained from medical record)
* For Clinically Stable Cohort: Clinically stable: free of any acute illness for >14 days
* For Clinically Stable Cohort: Must have performed spirometry for clinical purposes at that clinical visit
* For Clinically Stable Cohort: Must have a sputum culture sent to the clinical lab for clinical purposes at the time of the study visit
* For Clinically Stable Cohort: Have not been prescribed any new systemic antibiotics for the 14 days prior to enrollment
* For Exacerbation/IV Antibiotics Cohort: One copy of F508del
* For Exacerbation/IV Antibiotics Cohort: Must have a doctor defined pulmonary exacerbation requiring treatment with IV antibiotics
* For Exacerbation/IV Antibiotics Cohort: Must have performed spirometry for clinical purposes within 72 hours of initiating IV antibiotics and within 72 hours of completing IV antibiotics
* For Exacerbation/IV Antibiotics Cohort: Must have a sputum culture sent to the clinical lab for clinical purposes within 72 hours of admission

Exclusion Criteria:

* For Both Cohorts: Pregnancy (based on self-report)
* For Both Cohorts: Co-infection with Burkholderia cepacia complex organisms
* For Both Cohorts: Any condition that in the opinion of the subject or the subject's managing physician that would compromise that individuals ability to participate in these studies
* For Both Cohorts: Inability to tolerate the study procedures

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients seen in the cystic fibrosis outpatient clinic (Clinically Stable Cohort) and inpatient unit (Exacerbation/IV Antibiotics Cohort) of Cystic Fibrosis Center in Cleveland, OH (Rainbow Babies and Children's Hospital/University Hospitals Case Medical Center)
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2014-02; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James F. Chmiel, MD, MPH, Principal Investigator — Rainbow Babies and Children's Hospital
Locations (1):
- Rainbow Babies and Children's Hospital, Cleveland, Ohio, United States

REFERENCES:
- [Background] Chmiel JF, Berger M, Konstan MW. The role of inflammation in the pathophysiology of CF lung disease. Clin Rev Allergy Immunol. 2002 Aug;23(1):5-27. doi: 10.1385/CRIAI:23:1:005. PMID 12162106
- [Background] Lands LC, Stanojevic S. Oral non-steroidal anti-inflammatory drug therapy for lung disease in cystic fibrosis. Cochrane Database Syst Rev. 2013 Jun 13;(6):CD001505. doi: 10.1002/14651858.CD001505.pub3. PMID 23765216
- [Background] Flume PA, O'Sullivan BP, Robinson KA, Goss CH, Mogayzel PJ Jr, Willey-Courand DB, Bujan J, Finder J, Lester M, Quittell L, Rosenblatt R, Vender RL, Hazle L, Sabadosa K, Marshall B; Cystic Fibrosis Foundation, Pulmonary Therapies Committee. Cystic fibrosis pulmonary guidelines: chronic medications for maintenance of lung health. Am J Respir Crit Care Med. 2007 Nov 15;176(10):957-69. doi: 10.1164/rccm.200705-664OC. Epub 2007 Aug 29. PMID 17761616
- [Background] Oermann CM, Sockrider MM, Konstan MW. The use of anti-inflammatory medications in cystic fibrosis: trends and physician attitudes. Chest. 1999 Apr;115(4):1053-8. doi: 10.1378/chest.115.4.1053. PMID 10208207
- [Background] Konstan MW. Ibuprofen therapy for cystic fibrosis lung disease: revisited. Curr Opin Pulm Med. 2008 Nov;14(6):567-73. doi: 10.1097/MCP.0b013e32831311e8. PMID 18812834
- [Background] Konstan MW, Byard PJ, Hoppel CL, Davis PB. Effect of high-dose ibuprofen in patients with cystic fibrosis. N Engl J Med. 1995 Mar 30;332(13):848-54. doi: 10.1056/NEJM199503303321303. PMID 7503838
- [Background] Konstan MW, Schluchter MD, Xue W, Davis PB. Clinical use of Ibuprofen is associated with slower FEV1 decline in children with cystic fibrosis. Am J Respir Crit Care Med. 2007 Dec 1;176(11):1084-9. doi: 10.1164/rccm.200702-181OC. Epub 2007 Sep 13. PMID 17872492
- [Background] Chmiel JF, Konstan MW. Inflammation and anti-inflammatory therapies for cystic fibrosis. Clin Chest Med. 2007 Jun;28(2):331-46. doi: 10.1016/j.ccm.2007.02.002. PMID 17467552
- [Background] Taylor PR, Roy S, Leal SM Jr, Sun Y, Howell SJ, Cobb BA, Li X, Pearlman E. Activation of neutrophils by autocrine IL-17A-IL-17RC interactions during fungal infection is regulated by IL-6, IL-23, RORgammat and dectin-2. Nat Immunol. 2014 Feb;15(2):143-51. doi: 10.1038/ni.2797. Epub 2013 Dec 22. PMID 24362892

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Clinically Stable | Exacerbation
Started | 3 | 11
Completed | 3 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Clinically Stable | Exacerbation | Total
Number analyzed (Participants) | 3 | 11 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 11 | 14
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 6 | 7
  Male | 2 | 5 | 7
Region of Enrollment [Number; unit: participants]
  United States | 3 | 11 | 14

OUTCOME MEASURES:

1. Primary Outcome: Change in Sputum IL-17 Neutrophils
Description: In the Exacerbation/IV Antibiotics Cohort--Subjects will serve as their own controls. The percentage of neutrophils (in sputum) positive for IL-17 was determined by flow cytometry for each subject at the beginning and end of treatment for a pulmonary exacerbation. Sputum IL-17 neutrophil counts will be compared to the change in lung function (FEV1) as determined by spirometry (American Thoracic Society standards).
Time Frame: End of Treatment, two weeks. Samples will be obtained from each study volunteer at the beginning of IV antibiotic treatment and at the completion of antibiotic treatment for a pulmonary exacerbation
Population: Regarding "Clinically Stable" Arm: Because very few neutrophils at the end of treatment for a pulmonary exacerbation were positive for IL-17, it was determined not to undertake studies examining sputum neutrophils during periods of clinical stability.
Measure: Mean (Standard Deviation); unit: % of neutrophils positive for IL-17
Groups:
- Begining of Exacerbation: Study volunteer at the beginning of IV antibiotic treatment for a pulmonary exacerbation
- End of Exacerbation: Study volunteer at the completion of 2 weeks IV antibiotic treatment for a pulmonary exacerbation
Arm/Group | Begining of Exacerbation | End of Exacerbation
Number analyzed (Participants) | 11 | 11
% of neutrophils positive for IL-17 | 55 (23) | 4 (9)

2. Secondary Outcome: Sputum Inflammatory Mediators: IL-1β, IL-6, IL-8, IL-17A, TGF-β, TNF-α, and Neutrophil Elastase
Description: In the Clinically Stable Cohort--Measurement of sputum inflammatory mediators: IL-1β, IL-6, IL-8, IL-17A, TGF-β, TNF-α, and neutrophil elastase
Time Frame: Samples will be obtained at one outpatient clinic visit during the next calendar year
Population: Data not collected and will never be analyzed.
Groups:
- Clinically Stable Cohort: Clinically stable subjects
Arm/Group | Clinically Stable Cohort
Number analyzed (Participants) | 0

3. Secondary Outcome: Sputum Inflammatory Mediators: IL-1β, IL-6, IL-8, IL-17A, and Neutrophil Elastase
Description: In the Exacerbation/IV Antibiotics Cohort--Measurement of sputum inflammatory mediators by multiplex assay for IL-1β, IL-6, IL-8, and IL-17A. Neutrophil elastase determined by colorimetric assay. Measurements at the beginning of IV antibiotic treatment and after 2 weeks antibiotic treatment for a pulmonary exacerbation
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Begining of Exacerbation | End of Exacerbation
Number analyzed (Participants) | 11 | 11
pg/ml
  IL-1b (pg/ml) | 2313 (1452) | 757 (782)
  IL-6 (pg/ml) | 53 (26) | 37 (17)
  IL-8 (pg/ml) | 5785 (859) | 3428 (2604)
  IL-17 (pg/ml) | 302 (185) | 147 (152)
  Neutrophil elastase activity (pg/ml) | 195 (45) | 53 (45)

ADVERSE EVENTS:
Arm/Group | Clinically Stable | Exacerbation
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/11
Other Adverse Events (participants affected / at risk) | 0/3 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No